CLINICAL TRIAL: NCT02862314
Title: PROcalcitonin Pneumonia / Pneumonitis Associated With ASPIration
Acronym: PROPASPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2013/213
Record Dates: First submitted 2016-07-29; First posted 2016-08-11 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2020-05

CONDITIONS: Inhalation Pneumonia
Keywords: Procalcitonin
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Blood Specimen Collection

ARMS (2):
- procalcitonin group (Experimental): The procalcitonin concentration is measured at inclusion.
  Interventions: Biological: Blood sample
- control group (No Intervention): Concentrations of procalcitonin are not measured. .

INTERVENTIONS:
Biological: Blood sample
  Arms: procalcitonin group

SUMMARY:
There is actually no consensus in place defining for which patients with suspected inhalation pneumonia antibiotic treatment should be initiated and what the duration of this antibiotic treatment should be.

This absence of recommendations results in excessive use of antibiotics, in emergence of multi-resistant strains and increase of costs. Several studies have been performed investigating antibiotic treatment based on procalcitonin values and have demonstrated a decreased use of antibiotics without change in mortality rates, in duration of hospitalization, in occurrence of super-infections or in infection relapse rate. Of the studies performed in an intensive care setting, none has specifically studied inhalation pneumonia.

The objective of this study is to determine whether use of a decisional algorithm based on procalcitonin values allows reducing antibiotics exposure in patients who are intubated because of coma in comparison with standard care according to actual guidelines and clinical experience with respect to ventilator-acquired pneumonia.

The study has a prospective, multi-centre, comparative, randomized, open design. It is a superiority study, with as primary parameter the duration of antibiotic therapy during the first 15 days after admission in the intensive care unit (ICU).

Patients can be included in this study if they are intubated for coma (Glasgow Coma Scale (GCS) ≤ 8) within 48 hours following admission to the hospital and with a foreseen duration of ventilation exceeding 48 hours.

There will be two treatment groups, stratified by centre and randomised in blocs of 4: one group for which treatment initiation and discontinuation will be guided by a procalcitonin-based decisional algorithm and a control group to whom antibiotics will be administered according to the standard protocols of each participating centre.

Based on an estimated duration of antibiotic treatment of 6.2 days, a risk -significance α level- of 5%, a power of 90% and a reduction of antibiotic treatment duration of 25% in the treatment arm guided by procalcitonin values, the number of patients to be included is 83 per treatment arm. Taking into account a loss of 10% for patients lost to follow-up, 166 patients should be included.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older,
* have undergone oro-tracheal intubation for a coma (Glasgow Coma Score below or equal to 8),
* with mechanical ventilation initiated in the first 48 hours following hospital admission

Exclusion Criteria:

* pregnancy,
* patients under legal custody,
* patients without health insurance,
* patients included in another interventional clinical study involving infections or antibiotics and having the same primary parameter,
* moribund patients,
* situation in which the procalcitonin concentration could be increased without correlation to an infectious process (poly-traumatised patients,
* surgical interventions within the last 4 days,
* cardiorespiratory arrest,
* administration of anti-thymocyte globulin,
* immunodepressed patients (bone marrow transplant patients, patients with severe neutropenia),
* patients with an absolute indication for administration of antibiotics at the moment of ICU admission (meningitis, pneumonia) or a chronic infection for which long-term antibiotic treatment is necessary (endocarditis, osteo-articular infections, mediastinitis, deep abscesses, pneumocystis infection, toxoplasmosis, tuberculosis)
* patients with haemodynamic instability of septic origin or a respiratory insufficiency (defined by a ratio Pa02/Fi02 ≤ 200 mmHg and PEP ≥ 5 cmH2O)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
the duration of antibiotic treatment | during the first 15 days following admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Gilles CAPELLIER, MDPH, Principal Investigator — Centre hospitalier régional universitaire de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

REFERENCES:
- [Derived] Labro G, Aptel F, Puyraveau M, Paillot J, Pili Floury S, Merdji H, Helms J, Piton G, Ecarnot F, Kuteifan K, Quenot JP, Capellier G; PROPASPI (PROcalcitonin Pneumonia/pneumonitis Associated with ASPIration) trial investigators. Impact on antimicrobial consumption of procalcitonin-guided antibiotic therapy for pneumonia/pneumonitis associated with aspiration in comatose mechanically ventilated patients: a multicenter, randomized controlled study. Ann Intensive Care. 2021 Oct 12;11(1):145. doi: 10.1186/s13613-021-00931-4. PMID 34636974